CLINICAL TRIAL: NCT00642265
Title: The Treatment of Displaced, Midshaft Clavicular Fractures: Operative vs Conservative. A Prospected, Randomized Study
Brief Title: The Treatment of Clavicular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: AZ Sint-Jan AV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007/573
Record Dates: First submitted 2008-03-14; First posted 2008-03-25 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Displaced, Midshaft Clavicular Fractures
MeSH Terms: interventions — Fracture Fixation, Internal; Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): operative treatment
  Interventions: Procedure: osteosynthesis
- 2 (Active Comparator): conservative treatment
  Interventions: Other: sling

INTERVENTIONS:
Procedure: osteosynthesis — operative treatment
  Arms: 1
Other: sling — conservative treatment
  Arms: 2

SUMMARY:
Patients with a displaced, shortened, midshaft clavicular fracture are randomized in two groups: conservative or operative treatment. The conservative arm is treated with a sling for 6 weeks. The operative arm is treated with osteosynthesis, within 2 weeks.

Patients are clinically and radiologically evaluated during 1 year. A economical analysis is also done.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 year
* 100% displaced midshaft clavicular fracture
* shortening

  * male: 18mm
  * female: 14mm

Exclusion Criteria:

* pregnancy
* pathological fracture
* open fracture
* history of frozen shoulder
* ipsilateral fracture of shoulder or scapula
* neurovascular injury
* contraindication to anaesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-05-27 (Actual); Study Completion 2009-05-27 (Actual)

PRIMARY OUTCOMES:
Union | 1 year
Functionality | 1 year

SECONDARY OUTCOMES:
Complications | 1 year
Time to heal | 1 year
Cost | 1 year
Relation with medication | 1 year
Relation with smoking | 1 year
Relation with job | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lieven De Wilde, MD, PhD, Principal Investigator — University Hospital, Ghent; Bart Berghs, MD, Principal Investigator — AZ Sint-Jan AV; Pieter-Jan Vandekerckhove, MD, Principal Investigator — Sint-Andriesziekenhuis Tielt; J. Van Den Daele, MD, Principal Investigator — Stedelijk Ziekenhuis Roeselare; J. Vanonverschelde, MD, Principal Investigator — Stedelijk Ziekenhuis Aalst; G. Vandendriessche, MD, Principal Investigator — Jan Palfijnziekenhuis Ghent
Locations (6):
- Belgium (6):
  - Stedelijk Ziekenhuis Aalst, Aalst
  - AZ Sint Jan-Brugge, Bruges
  - Jan Palfijnziekenhuis, Ghent
  - University Hospital Ghent, Ghent
  - Stedelijk Ziekenhuis Roeselare, Roeselare
  - Sint-Andries Ziekenhuis, Tielt

REFERENCES:
- See also: Related Info — http://www.uzgent.be